CLINICAL TRIAL: NCT00104936
Title: Observation Versus Conventional-Fractionated Radiotherapy or Radiosurgery After Non-radical Surgery for Benign Intracranial Meningiomas: A Phase III Study
Brief Title: Radiotherapy or Radiosurgery Compared With Observation Alone in Treating Patients With Newly Diagnosed, Benign Meningioma That Has Been Partially Removed by Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-26021 -22021; EORTC-26021; EORTC-22021; CAN-NCIC-EORTC-26021
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult grade I meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Chemotherapy, Adjuvant; Radiotherapy; Radiosurgery

INTERVENTIONS:
Procedure: adjuvant therapy
Radiation: radiation therapy
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Giving radiation therapy or radiosurgery after surgery may kill any remaining tumor cells. It is not yet known whether radiation therapy or radiosurgery is more effective than observation alone in treating benign meningioma.

PURPOSE: This randomized phase III trial is studying radiation therapy or radiosurgery to see how well they work compared to observation alone in treating patients with newly diagnosed, benign meningioma that has been partially removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of patients with newly diagnosed, incompletely resected, benign intracranial grade I meningioma treated with adjuvant conventional fractionated radiotherapy or radiosurgery vs observation only.

Secondary

* Compare the quality of life of patients treated with these regimens.
* Compare overall survival of patients treated with these regimens.
* Compare the incidence of a second surgery in patients treated with these regimens.
* Compare the incidence of acute and long-term neurotoxicity in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to post-surgery MRI staging (3 vs 4 vs 5), skull base location (yes vs no), age (< 60 vs ≥ 60), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo observation only.
* Arm II: Within 4-7 months after surgery, patients undergo conventional fractionated radiotherapy once daily, 5 days a week for 6 weeks OR a single treatment of high-dose radiosurgery in the absence of unacceptable toxicity.

Quality of life is assessed at baseline, at 6 months after randomization, and then annually thereafter.

After completion of study treatment, patients are followed at 3 and 6 months after randomization and then annually thereafter.

PROJECTED ACCRUAL: A total of 478 patients (239 per treatment arm) will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed benign intracranial meningioma

  * WHO grade I
  * Any location except orbital meningioma
* Mitotic index < 4 (total counts per 10 high-power field) AND MIB-1 labeling index < 4%
* The following histologies are not allowed (i.e., WHO grade II or III):

  * Atypical
  * Clear cell
  * Choroid
  * Rhabdoid
  * Papillary
  * Anaplastic
* Must have undergone non-radical resection* within the past 7 months

  * Post-operative MRI (performed 4 months after surgery) demonstrating stages 3, 4, or 5 NOTE: *Biopsy only is considered non-radical resection and may be classified as stage 4 or 5 according to tumor volume
* No brain invasion
* No hemangiopericytoma
* No fibrous dysplasia or intra-osseous meningioma
* No multiple meningiomas or meningiomatosis
* Not part of neurofibromatosis type II

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No serious congestive heart failure

Other

* HIV negative
* No other malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No other disease that would preclude 5-year follow up after study completion
* No psychological, familial, sociological, or geographical condition that would preclude study compliance or study follow up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the meninges or brain that would preclude study treatment

Surgery

* See Disease Characteristics

Other

* No prior randomization to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-12; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Quality of life
Overall survival
Incidence of a second surgery
Acute neurotoxicity
Long-term neurotoxicity

CONTACTS AND LOCATIONS:
Overall Officials: John G. Wolbers, MD, PhD, Study Chair — University Medical Center Rotterdam at Erasmus Medical Center; Raymond Miralbell, MD, Study Chair — Hopital Cantonal Universitaire de Geneve; Rolando F. Del Maestro, MD, PhD, Study Chair — Montreal Neurological Institute and Hospital; Luis Souhami, MD, Study Chair — McGill Cancer Centre at McGill University
Locations (4):
- University Hospital Schleswig-Holstein - Kiel Campus, Kiel, Germany
- Netherlands (2):
  - Radiotherapeutisch Instituut-(Riso), Deventer
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
- Hopital Cantonal Universitaire de Geneve, Geneva, Switzerland